CLINICAL TRIAL: NCT06440915
Title: Study on Theraputic Drug Monitoring and Phamacokinetics of Isavuconazole in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Principal Investigator, Juan Wu, PhD, Principal Investigator, Shanghai Children's Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YJK-001
Record Dates: First submitted 2024-05-20; First posted 2024-06-04 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Aspergillosis Invasive; Mucormycosis
MeSH Terms: conditions — Mucormycosis | interventions — isavuconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isavuconazole group (Other): Theraputic drug monitoring
  Interventions: Other: Theraputic drug monitoring; Drug: Isavuconazole

INTERVENTIONS:
Other: Theraputic drug monitoring — High Performance Liquid Chromatography (HPLC) is used to determine the plasma concentrations of isavuconazole
Drug: Isavuconazole — Isavuconazole

SUMMARY:
The goal of this clinical trial is to learn the plasma concentration of isavuconazole in pediatric patients. It will also learn about the relationship of isavuconazole plasma concentrations to efficacy and safety in pediatric patients. The main questions it aims to answer are:

What is the plasma concentration after using isavuconazole in pediatric patients? What is the effective range of plasma concentration of isavuconazole in pediatric patients? What is the safe range of plasma concentration of isavuconazole in pediatric patients? Researchers will measure the plasma concentration of isavuconazole to see whether it is appropriate.

Participants will:

Take drug isavuconazole as prescribed by the doctor;

1mL of blood is drawn 30min before the next dose.

DETAILED DESCRIPTION:
Objectives of Study:

Main objective: To monitor the plasma concentration of isavuconazole in children, and to study the pharmacokinetic characteristics of isavuconazole in children, so as to provide basis for the optimization of individualized drug administration.

Secondary objective: To evaluate the relevance of isavuconazole plasma concentrations to efficacy and safety in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who intend to take isavuconazole for the treatment of invasive mycosis;
* Aged 0-18 years, gender unlimited;
* The subject and his/her guardian are willing to comply with the procedures and operations specified in the study protocol;
* The guardian of the subject and the subject of independent informed age are willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

* The subject is known to be allergic to any azole antifungal therapy or other ingredients contained in the study drug;
* The researcher believes that the condition of the child may interfere with study participation or other inappropriate conditions.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of isavuconazole | 30 minutes before next dosing
  High Performance Liquid Chromatography is used to determine the plasma concentrations of isavuconazole

SECONDARY OUTCOMES:
Treatment success rates for IMI | 6 months
  Percentage of patients who were assessed by the study physician as clinically cured and improved
AE and SAE | 6 months
  Number and percentage of AE and SAE

CONTACTS AND LOCATIONS:
Overall Officials: Juan Wu, PhD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Date of sharing: after publication of the study results; Way of sharing: Contact the investigator for request
Supporting Information: Study Protocol, CSR
Time Frame: After publication of the study results
Access Criteria: Contact the investigator for request